CLINICAL TRIAL: NCT03135093
Title: Assessing Pathological Synergies of Upper Limb Function and the Relationship to Visuospatial Exploration After Stroke
Brief Title: Upper Limb Function and Visuospatial Exploration After Stroke
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-02075
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: synergies; upper limb; vision
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke subjects
  Interventions: Other: No intervention
- Healthy subjects
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
This project is a cross-sectional, observational mono-center study with prospective data collecting.

This study aims to further explore quality of upper limb movement in relation to characteristics of visuospatial exploration in stroke subjects and healthy subjects by a applying comprehensive measurements of clinical scales and kinematic data in capacity- and performance-based activities. The results will contribute to assessing and monitoring quality of upper limb movements and visuospatial attention and their relationship.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 18 years and older with chronic ischemic stroke (> 6 month) restricted to one hemisphere (confirmed by CT/MRI)
* With impairments in upper limb function and at least partial ability to lift the arm against gravity, flex and extend the fingers
* Without relevant pre-existing limitations in arm and hand function (orthopaedic, muscular, neurologic)
* Written informed consent after participants's information

Exclusion Criteria:

* Increased muscle tone in the upper limb with limited rang of motion
* Severe sensory deficits in the upper limb
* Clinically significant concomitant disease (affecting the upper limb or impaired vision, e.g. due to glaucoma etc.)
* Contraindications on ethical grounds (vulnerable persons)
* Known or suspected non-compliance, drug or alcohol abuse
* Severe communication or cognitive deficits, that cause inability to follow the procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke subjects
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Upper limb movement quality | One day
  Fugl-Meyer Assessment of the upper extremity (FMA-UE), kinematic data (e.g. joint angles, hand workspace)
Visuospatial exploration | One day
  Eye-tracking data (e.g. area of interest, eye movements: saccades, fixations) and to rule out stroke-related deficits of visuospatial attention, clinical tests

CONTACTS AND LOCATIONS:
Locations (1):
- cereneo Schweiz AG, Vitznau, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The anonymized project data will be shared within the partners of the European Horizon2020 - SoftPro (No.688857) project.

REFERENCES:
- [Derived] Schwarz A, Bhagubai MMC, Nies SHG, Held JPO, Veltink PH, Buurke JH, Luft AR. Characterization of stroke-related upper limb motor impairments across various upper limb activities by use of kinematic core set measures. J Neuroeng Rehabil. 2022 Jan 12;19(1):2. doi: 10.1186/s12984-021-00979-0. PMID 35016694
- [Derived] Schwarz A, Veerbeek JM, Held JPO, Buurke JH, Luft AR. Measures of Interjoint Coordination Post-stroke Across Different Upper Limb Movement Tasks. Front Bioeng Biotechnol. 2021 Jan 28;8:620805. doi: 10.3389/fbioe.2020.620805. eCollection 2020. PMID 33585418